CLINICAL TRIAL: NCT00218361
Title: Biobehavioral Study of Opioid Drug Seeking Behavior: Study 2
Brief Title: Effects of Post-Session Supplemental Hydromorphone on Drug Seeking Behavior in Opioid Dependent Individuals
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark Greenwald, PhD, Principal Investigator, Wayne State University
Other Study IDs: NIDA-15462-2; R01DA015462 (NIH); R01-15462-2; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Heroin Dependence; Opioid-Related Disorders
Keywords: Behavioral economics; Drug self administration; Opioid
MeSH Terms: conditions — Heroin Dependence; Opioid-Related Disorders | interventions — Hydromorphone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood

INTERVENTIONS:
Drug: Hydromorphone

SUMMARY:
The purpose of this study is to determine whether knowledge of post-session hydromorphone (HYD) availability reduces drug seeking behavior in heroin dependent individuals.

DETAILED DESCRIPTION:
Drug dependence is often characterized by severe drug seeking behavior. Learning to understand, predict, and control this maladaptive choice behavior may lead to improved prevention and treatment strategies. HYD is a drug that is currently used as a cough suppressant and to relieve pain. The purpose of this study is to determine the extent to which opioid drug seeking behavior by heroin dependent individuals can be reduced by environmental factors, including supplemental opioid drug availability, drug price, and alternative non-drug reinforcers. Specifically, this study will determine whether knowledge of post-session HYD availability influences drug seeking behavior in heroin dependent individuals, who are maintained on buprenorphine during their participation.

Participants in this observational study will take part in multiple trials in which they have the opportunity to choose either HYD or money. On the first two experimental days, prior to choice sessions, participants will receive a sample of the drug doses that can be chosen. During test sessions, participants will have 12 opportunities to choose either drug or money. Participants will use a computer to earn choices. Respiration rate, oxygen saturation, heart rate, and blood pressure will be monitored throughout choice trials. Supplemental HYD will be made available following some choice sessions. Self-report questionnaires will be completed at different times during the study. Participants will be maintained on buprenorphine throughout the study, with a minimum 2-week lead before the experiment, and a fixed 3-week detoxification after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Opioid dependent, as determined by the structured clinical interview for DSM-IV (SCID) and Addiction Severity Index (ASI)
* Positive urine test for opiates
* Willing to use an adequate form of contraception for the duration of the study
* Reads and writes English

Exclusion Criteria:

* Psychiatric illness, as determined by the DSM-IV criteria
* History of or current neurological disease, including structural abnormalities, seizures, infection, peripheral neuropathy, and head traumas
* History of cardiovascular disease, myocardial infarction, chest pain, or edema
* Systolic blood pressure greater than 160 mm Hg or less than 95 mm Hg; PR diastolic blood pressure greater than 95 mm Hg
* Pulmonary disease, including obstructive pulmonary disease, cor pulmonale, tuberculosis, and asthma
* Systemic disease (e.g., endocrinopathies, liver or kidney failure, myxedema, hypothyroidism, Addison's disease, autoimmune disease)
* Current alcohol or sedative drug dependence
* Pregnant or breastfeeding
* Currently receiving treatment for opioid dependence
* Known phobia of injections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Heroin dependent research volunteers
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Mark Greenwald, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University, Detroit, Michigan, United States

REFERENCES:
- [Derived] Woodcock EA, Lundahl LH, Burmeister M, Greenwald MK. Functional mu opioid receptor polymorphism (OPRM1 A(118) G) associated with heroin use outcomes in Caucasian males: A pilot study. Am J Addict. 2015 Jun;24(4):329-35. doi: 10.1111/ajad.12187. Epub 2015 Apr 24. PMID 25911999
- [Derived] Stoltman JJ, Woodcock EA, Lister JJ, Greenwald MK, Lundahl LH. Exploration of the telescoping effect among not-in-treatment, intensive heroin-using research volunteers. Drug Alcohol Depend. 2015 Mar 1;148:217-20. doi: 10.1016/j.drugalcdep.2015.01.010. Epub 2015 Jan 19. PMID 25630964
- [Derived] Greenwald MK, Steinmiller CL, Sliwerska E, Lundahl L, Burmeister M. BDNF Val(66)Met genotype is associated with drug-seeking phenotypes in heroin-dependent individuals: a pilot study. Addict Biol. 2013 Sep;18(5):836-45. doi: 10.1111/j.1369-1600.2011.00431.x. Epub 2012 Feb 16. PMID 22339949